CLINICAL TRIAL: NCT02436226
Title: Use of Low Dose of Human Chorionic Gonadotropin During Ovulation Induction With Clomiphene Citrate in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome
Brief Title: Use of Low Dose of HCG During Ovulation Induction With CC in Women With CC Resistant PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT1
Record Dates: First submitted 2015-05-02; First posted 2015-05-06 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: PCOS; Clomiphene citrate resistant; HCG
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Clomiphene; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene citrate-HCG group (Active Comparator): Women will receive clomiphene citrate and human chorionic gonadotropin (HCG)
  Interventions: Drug: Clomiphene citrate and Human chorionic gonadotropin (HCG)
- Clomiphene citrate group (Active Comparator): Women will receive clomiphene citrate alone
  Interventions: Drug: Clomiphene citrate

INTERVENTIONS:
Drug: Clomiphene citrate and Human chorionic gonadotropin (HCG) — Women will receive clomiphene citrate (150 mg/day for 5 consecutive days from day 2 of cycle) and HCG (200 IU/day SC from day 7 of cycle)
  Other Names: Clomid and Choriomon
  Arms: Clomiphene citrate-HCG group
Drug: Clomiphene citrate — Women will receive clomiphene citrate (150 mg/day for 5 consecutive days from day 2 of cycle)
  Other Names: Clomid
  Arms: Clomiphene citrate group

SUMMARY:
The purpose of this study is to evaluate the effect of administration of low dose of human chorionic gonadotropin (HCG) after use of clomiphene citrate (CC) for induction of ovulation in infertile women having CC resistant polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; CC-HCG group and CC group. Women in the CC-HCG group will receive CC (150 mg/day for 5 consecutive days from day 2 of cycle) and HCG (200 IU/day SC from day 7 of cycle). Women in the CC group will receive CC alone (150 mg/day for 5 consecutive days from day 2 of cycle). Transvaginal sonography (TVS) scan will be performed regularly for monitoring of follicular growth (folliculometry); starting from day 10 of the stimulation cycle and repeated every 2-3 days. When there will be at least one follicle ≥ 18 mm in diameter, final oocyte maturation will be induced by intramuscular administration of 10000 IU of HCG and timed intercourse will be advised. If there will be no follicle ≥ 12 mm by day 16 of the cycle, monitoring of follicular growth will be discontinued and the cycle will be presumed to be anovulatory. Ovulation will be documented by TVS scan one week after triggering of oocyte maturation and will be confirmed by assessing the midluteal serum progesterone level. Each woman will be subjected to ovarian stimulation for a maximum of 3 consecutive cycles except if she gets pregnant in the first or second cycle

ELIGIBILITY:
Inclusion Criteria:

* Infertile lean women with PCOS as defined by the Rotterdam criteria.
* CC resistance (defined as failure of ovulation after receiving 150 mg/day of CC for 5 consecutive days per cycle, for at least 3 consecutive cycles).

Exclusion Criteria:

* Age < 20 or > 35 years.
* Presence of any infertility factor other than anovulatory PCOS.
* Previous history of ovarian surgery or surgical removal of one ovary.
* Previous exposure to cytotoxic drugs or pelvic irradiation.
* Oral hypoglycemic or hormonal therapy either currently or in the preceding 3 months.
* Metabolic or hormonal abnormalities.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 3 months
  Number of ovulatory cycles divided by the number of stimulation cycles

SECONDARY OUTCOMES:
Number of ovarian follicles ≥ 18 mm on day of triggering of oocyte maturation | 3 months
  Number of ovarian follicles ≥ 18 mm by TVS on day of triggering of oocyte maturation
Endometrial thickness on day of triggering of oocyte maturation | 3 months
  Endometrial thickness by Transvaginal sonography (TVS) scan on day of triggering of oocyte maturation
Clinical pregnancy rate | 6-8 weeks gestational age
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 6-8 weeks gestational age) divided by the number of women
Incidence of early ovarian hyperstimulation syndrome (OHSS) | Within 9 days of final triggering of oocyte maturation
  Incidence of OHSS within 9 days of final triggering of oocyte maturation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Thabet, MD, Principal Investigator — Mansoura University; Khaled S Ismael, MD, Study Director — Mansoura University; Ahmed Ragab, MD, Study Director — Mansoura University; Maged R Elshamy, MD, Study Director — Mansoura University; Mohamed A Elnegery, MD, Study Director — Mansoura University; Hamed Youssef, MD, Study Director — Mansoura University; Mahmoud M Abdel-razik, MD, Study Director — Mansoura University; Mohamed S Abdelhafez, MD, Study Chair — Mansoura University
Locations (1):
- Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thabet M, Abdelhafez MS, Elshamy MR, Albahlol IA, Fayala E, Wageeh A, El-Zayadi AA, Bahgat NA, Mohammed SM, Mohamed AA, Awad MM, El-Menayyer A, El-Sherbiny M, Elsherbini DMA, Albarakati RG, Alshaikh ABA, Edris FE, Bushaqer NJ, Salama YGM, Abdel-Razik MM. Competence of Combined Low Dose of Human Chorionic Gonadotropin (HCG) and Clomiphene Citrate (CC) Versus Continued CC during Ovulation Induction in Women with CC-Resistant Polycystic Ovarian Syndrome: A Randomized Controlled Trial. Medicina (Kaunas). 2024 Aug 12;60(8):1300. doi: 10.3390/medicina60081300. PMID 39202581